CLINICAL TRIAL: NCT04360629
Title: Efficacy and Safety of Tranexamic Acid in Cytoreductive Surgery for Ovarian Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jun Zhang (Other)
Responsible Party: Sponsor-Investigator, Jun Zhang, Director of the department of anaesthesiology, Shanghai cancer center, Fudan University
Organization: Fudan University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: V1.0
Record Dates: First submitted 2020-04-22; First posted 2020-04-24 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Advanced Ovarian Cancer
MeSH Terms: interventions — Tranexamic Acid; Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- high dose TXA (Experimental): TXA will be given as a 20mg/kg bolus followed by infusion of 5mg/ kg/hr per our anesthesia protocol
  Interventions: Drug: Tranexamic Acid
- low dose TXA (Experimental): TXA will be given as a 10mg/kg bolus followed by infusion of 1mg/ kg/hr per our anesthesia protocol
  Interventions: Drug: Tranexamic Acid
- normal saline (Placebo Comparator): saline will be given as a 4ml/kg bolus followed by infusion of 1ml/ kg/hr per our anesthesia protocolprotocol4ml/kg
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: Tranexamic Acid — Tranexamic Acid will be given through central vein
  Arms: high dose TXA; low dose TXA
Drug: normal saline — normal saline will be given through central vein
  Arms: normal saline

SUMMARY:
Tranexamic acid has been used in surgery for more than 30 years. It's effect on reducing bleeding and blood transfusing has been demonstrated.

In our hospital, the amount of cytorsductive surgery for ovarian cancer is big. During the perioperation , bleeding probability is high, and the supply of blood products is limited. In order to reduce bleeding, we're planning to use tranexamic acid in the operations.

In this experiment, we will observe the efficacy of tranexamic acid in cytoreductive surgery for ovarian cancer, find the best dosage which can reach the desired effect, and the possible side-effect.

DETAILED DESCRIPTION:
We performed a single blind, prospective, randomised control trial (RCT) . The patients randomised assigned to three groups. Low dose TXA, high dose TXA or a placebo of IV saline which will be infused prior to skin incision in patients undergoing elective cytorsductive surgery for ovarian cancer .

Intraoperative blood loss will be estimated by the volume in the suction drains and by weighing the swabs. Postoperative blood loss will be estimated by the volume in the drains.

The other secondary outcomes will be inclued perioperation transfusion volume, thromboembolic complications, ICU length of stay (LOS), hospital LOS, adverse thrombogenic events within 30 days, 30-day all-cause readmission and so on.

ELIGIBILITY:
Inclusion Criteria:

1. sign the informed consent
2. Aged 20-70 years
3. ovarian cancer patients, staged IIIB - C or above

3) ASA I - II

Exclusion Criteria:

1. tranexamic acid allergy
2. pregnancy and lactation
3. only lymph node metastasise
4. history of mental disorder, immune system disorder
5. history of epilepsy, dyschromatopsia
6. arrhythmia
7. history of renal insufficiency
8. thrombosis related disease
9. Hb < 90 g/dL
10. using anticoagulant drugs (not including aspirin discontinuation 1 week
11. having participated in other clinical trials, or refusing to join the research.

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2020-06-03 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
operative and postoperative blood loss | up to 8 days
  the amount of bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Jun Zhang, PhD, Principal Investigator — Fudan University
Locations (1):
- Shanghai Cancer Center, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zakhari A, Sanders AP, Solnik MJ. Tranexamic acid in gynecologic surgery. Curr Med Res Opin. 2020 Mar;36(3):513-520. doi: 10.1080/03007995.2019.1708533. Epub 2020 Jan 6. PMID 31865770
- [Result] Kietpeerakool C, Supoken A, Laopaiboon M, Lumbiganon P. Effectiveness of tranexamic acid in reducing blood loss during cytoreductive surgery for advanced ovarian cancer. Cochrane Database Syst Rev. 2016 Jan 23;2016(1):CD011732. doi: 10.1002/14651858.CD011732.pub2. PMID 26801659
- [Result] Lundin ES, Johansson T, Zachrisson H, Leandersson U, Backman F, Falknas L, Kjolhede P. Single-dose tranexamic acid in advanced ovarian cancer surgery reduces blood loss and transfusions: double-blind placebo-controlled randomized multicenter study. Acta Obstet Gynecol Scand. 2014 Apr;93(4):335-44. doi: 10.1111/aogs.12333. Epub 2014 Feb 25. PMID 24428857
- [Result] Heyns M, Knight P, Steve AK, Yeung JK. A Single Preoperative Dose of Tranexamic Acid Reduces Perioperative Blood Loss: A Meta-analysis. Ann Surg. 2021 Jan 1;273(1):75-81. doi: 10.1097/SLA.0000000000003793. PMID 32224739
- [Derived] Yang X, Chai M, Xia L, He Z, Wu X, Zhang J. Intraoperative use of tranexamic acid to reduce blood loss during cytoreductive surgery for advanced ovarian cancer: A randomized controlled clinical trial. Acta Obstet Gynecol Scand. 2023 Jul;102(7):950-959. doi: 10.1111/aogs.14567. Epub 2023 Apr 7. PMID 37029431